CLINICAL TRIAL: NCT00276536
Title: Phase I Evaluation of Interferon-alpha-1b in Solid Tumors, Lymphoma or Myeloma
Brief Title: Interferon Alfa in Treating Patients With Stage IV Solid Tumors, Lymphoma, or Myeloma
Acronym: IFNa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-3575; P30CA043703 (NIH); CASE-CCF-3575 (Other: IRB)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Kidney Cancer; Lymphoma; Melanoma; Multiple Myeloma; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV melanoma; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Kidney Neoplasms; Lymphoma; Melanoma; Multiple Myeloma; Sarcoma | interventions — interferon-alfa-1b; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): IFN weekly
  Interventions: Biological: recombinant interferon alpha-1b; Drug: IFN

INTERVENTIONS:
Biological: recombinant interferon alpha-1b — interferon
  Other Names: Interferon
Drug: IFN — IFN daily
  Other Names: Interferon

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells and slow the growth of cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of interferon alfa in treating patients with stage IV solid tumors, lymphoma, or myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Confirm tolerance and safety of interferon alfa-1b (IFN-α1b) in patients with stage IV solid tumors, lymphoma, or myeloma.
* Determine the maximum tolerated dose (MTD) of IFN-α1b given daily by subcutaneous injection in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive interferon alfa-1b subcutaneously once daily for at least 1 month. Treatment continues for up to 12 months in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of interferon alfa-1b until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy, including, but not limited to, renal cell carcinoma, melanoma, Kaposi's sarcoma, breast carcinoma, lymphoma, myeloma, or tumors of endothelial origin

  * Stage IV disease
  * Refractory to standard therapy
* Measurable or evaluable disease

  * Evaluable disease can include clinically or radiographically nonmeasurable tumor or specific tumor markers
* Patients with prior solitary CNS metastasis allowed

  * Must have had prior definitive therapy ≥ 3 months previously
  * No requirement for glucocorticoids unless for physiologic replacement
* No multiple CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.3 times upper limit of normal (ULN) OR
* Creatinine clearance of 60 mL/min
* Bilirubin ≤ 1.3 times ULN
* AST ≤ 5 times ULN
* No pregnant or lactating women
* Fertile women and men, unless surgically sterile, must use effective contraception
* No history of serious cardiac arrhythmia or cardiac arrhythmia requiring treatment
* No congestive heart failure
* No angina pectoris
* No New York Heart Association class III or IV disease
* No other severe cardiovascular disease
* No known seizure disorder
* No known HIV or hepatitis B surface antigen positivity
* No active clinical infection requiring antibiotics within the past 7 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 months since prior interferon therapy and/or ≤ 400 million units of interferon
* At least 3 weeks since prior major surgery requiring general anesthesia
* At least 3 weeks since prior radiotherapy or chemotherapy
* Treatment with hormones or other chemotherapeutic agents may not be administered except for steroids given for preexisting adrenal failure or hormones administered for nondisease-related conditions (e.g., insulin for diabetes)
* No prior organ allograft
* No concurrent dexamethasone, other steroidal antiemetics, or anti-inflammatories
* No concurrent palliative radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Tolerance and safety as measured by any ≥ Grade IV granulocyte toxicity or any Grade III toxicity thought to be drug related at 1 week after each course | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ernest C. Borden, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States